CLINICAL TRIAL: NCT05323409
Title: Optimise: Improving Comprehensive Care of Cancer Patients With Comorbidities
Brief Title: Improving Comprehensive Care of Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Hoda Badr, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-49731
Record Dates: First submitted 2021-07-14; First posted 2022-04-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Gastrointestinal Cancer; Hematologic Cancer
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OPTIMISE (Experimental): OPTIMISE components to facilitate Patient self-management support are: 1) a bilingual oncology nurse navigator (ONN) and care coordination; 2) distress screening; 3) tailored comorbidity self-management action planning, 4) tailored survivorship action planning, and 5) surveillance reminders and follow-up. OPTIMISE components to facilitate provider decision support are: 1) when the initial referral is made, the ONN will send the PCP treatment plan summary (based on the ASCO treatment plan template) and standardized fact sheets on treatment toxicities; 2) throughout treatment, there will be bi-directional and structured communication between oncologist and PCP facilitated by the ONN; 3) The ONN will send the SCP to the PCP describing surveillance guidelines and summary of late effects. Finally, OPTIMISE will adopt a risk-stratified shared care model of post-treatment survivorship care.
  Interventions: Behavioral: OPTIMISE
- Usual Medical Care (UMC) (No Intervention): UMC consists of standard oncologic care from point of diagnosis. Cancer patients with comorbidities are encouraged by their oncologist to follow up with their PCP regarding comorbidity management but no formal referral process is in place. At the end of cancer treatment (with standard, definitive therapies), patients meet with a nurse (Survivorship Nurse Practitioner, NP) to review the SCP, which is based on ASCO templates and populated from the EHR. The Survivorship NP also reviews therapies received, recommended surveillance, common late effects, and recommended lifestyle behaviors. Patients are given a printed copy of the SCP and are encouraged to share this information with their PCP. Cancer surveillance follows the traditional oncologist led model regardless of patient risk for recurrence.

INTERVENTIONS:
Behavioral: OPTIMISE — OPTIMISE is a multilevel intervention that seeks to improve patient activation for comorbidity self-management during cancer treatment and coordination of care between oncologists and primary care physicians from point of diagnosis through the first year of post-treatment survivorship.
  Arms: OPTIMISE

SUMMARY:
Cancer survivors have unique healthcare needs, including managing serious late effects, ongoing surveillance, lifestyle modifications to reduce second cancer risk, and psychosocial support. Nearly 70% of survivors have at least one comorbid chronic condition in addition to cancer, which complicates the delivery of quality cancer care. Medically underserved patients, who bear the highest burden of multiple chronic conditions, are at increased risk for poor outcomes during and after cancer treatment. Enhancing communication and collaboration between oncologists and primary care providers (PCPs) could improve health outcomes and care transitions for these patients, who often lack healthcare knowledge and access to supportive care.

This study evaluates a novel shared care model for cancer survivors with chronic comorbidities, called OPTIMISE (Oncology-Primary Care Partnership to Improve Comprehensive Survivorship Care), in the largest safety-net healthcare system in Houston, Texas. Three hundred newly diagnosed breast, gastrointestinal, and hematological cancer patients being treated with curative intent and having comorbidities requiring ongoing management will be randomized to either OPTIMISE or Usual Medical Care (UMC). UMC patients will receive cancer treatment directed by their oncologist, a survivorship care plan (SCP) at the end of active treatment, and surveillance visits based on national guidelines.

OPTIMISE patients will: 1) have an oncology nurse navigator assigned to their care team at diagnosis to facilitate oncologist-PCP communication; 2) receive coordinated care between their oncologist and PCP throughout cancer treatment and surveillance, facilitated by structured communication and referral processes; 3) receive an SCP that incorporates comorbidity management; and 4) follow a risk-stratified shared care model where some routine oncologist follow-up visits are replaced by PCP visits. Aim 1a evaluates OPTIMISE's impact on patient chronic disease self-management (primary outcome) and quality of life (secondary outcome). Aim 1b explores OPTIMISE's effects on healthcare use and patient unmet needs during and after treatment. Aim 2 examines OPTIMISE's impact on oncologist and PCP attitudes and care coordination. Aim 3 elucidates patient- and system-level factors influencing implementation outcomes. If effective, OPTIMISE could expand to other cancers and enhance care transitions in various medical settings.

DETAILED DESCRIPTION:
Design Overview. This is a randomized controlled trial of a consecutive sample of 300 medically underserved breast, GI, and hematological cancer patients with comorbidities recruited from Harris Health Ben Taub Hospital and Smith Clinic. Randomization will divide patients into two groups. The first is those receiving UMC.

The second is those receiving OPTIMISE. Grounded by the Collaborative Chronic Care Model (CCM), OPTIMISE targets patients, providers, and systems of care. Key components are 1) a bilingual ONN, 2) culturally tailored self management action planning, 3) a referral schedule and structured communication between oncologists and PCPs, 3) an EHR generated SCP, and 4) a risk stratified shared care model for cancer surveillance. Patients in both arms will complete surveys at baseline (cancer treatment planning visit), during routine clinic visits at 2 and 4 months after cancer treatment initiation/study enrollment, the time of SCP delivery, and 3, 6, and 12 months after SCP delivery. Healthcare providers complete surveys upon enrollment and study completion. We will also interview patients and providers to understand experiences with comorbidity management and care transitions and identify individual and system barriers to future adoption, implementation, and sustainability of OPTIMISE. Recruitment and Baseline Assessment. Provider Recruitment. Before starting patient recruitment, the research assistant (RA) will consent oncologists and PCPs using a blanket consent. Reasons for refusal will be tracked. All providers will complete a short baseline survey to assess collaboration, satisfaction with comorbidity care management and care transitions. Patient Recruitment. The RC will approach potentially eligible patients during routine clinic visits, introduce the study, and obtain informed consent. Consenting patients will be asked to complete the baseline survey on tablet computers using REDCap in the waiting room. Surveys are brief (30 minutes) to minimize burden. As wait times are usually more than 1 hour, patients should have ample time to complete the survey. Patients will then be randomized to UMC or OPTIMISE. Patients who are randomized to OPTIMISE will be referred to a Harris Health PCP if they do not currently have one.

Study Arms. UMC consists of standard oncologic care from point of diagnosis. Cancer patients with comorbidities are encouraged by their oncologist to follow up with their PCP regarding comorbidity management but no formal referral process is in place. At the end of cancer directed treatment patients meet with a nurse (Survivorship Nurse Practitioner, NP) to review the SCP, which is populated from the electronic health record. The Survivorship NP also reviews therapies received, recommended surveillance, common late effects, and recommended lifestyle behaviors. Patients are given a printed copy of the SCP and are encouraged to share this information with their PCP. Cancer surveillance follows the traditional oncologist led model regardless of patient risk for recurrence. OPTIMISE seeks to improve comprehensive care and outcomes for underserved cancer patients with comorbidities from diagnosis to survivorship. It is based on IOM recommendations, our preliminary data, and the Collaborative Chronic Care Model (CCM). The CCM seeks to optimize 6 elements of care 1) self management support, 2) provider decision support, 3) use of clinical information systems, 4) delivery system redesign, 5) linkages to community resources, and 6) organizational support. OPTIMISE components organized by CCM elements are described below.

Patient Self management Support. ONN care coordination. The ONN will meet with the patient to 1) explain the navigator role, 2) answer questions about cancer treatment and next steps, and, 3) provide a resource list of hospital and community resources (e.g., counselors, translators) based on stated needs. The ONN will also coordinate a referral to a Harris Health PCP for comorbidity management. The ONN will follow up with the patient and PCP to ensure the visit occurs within 1 month of referral. Distress screening. At the initial oncology consult, patients will complete the NCCN Distress Thermometer and problem checklist. All distressed patients (scores greater than 5 out of 10) are referred to social work and receive a mental health resource list. For those receiving OPTIMISE, the ONN will additionally notify the PCP so causes of distress can be further explored and the patient connected to appropriate support resources. Culturally tailored comorbidity self management action planning. After the patients initial PCP consult, the ONN will review the PCPs progress notes in EPIC regarding the recommended comorbidity management plan. The ONN will send a memo to the PCP via his or her EPIC mailbox requesting clarifications as needed. Based on this, at the patients next routine oncology clinic visit, the ONN and patient will collaborate on a comorbidity self management action plan. A brief action planning approach will be employed whereby the patient identifies a specific, actionable self management goal (e.g., diet change, medication adherence), actions to work toward achieving the goal, possible barriers and solutions, where, how much, how often, and when the action will occur, and how and when the patient will self check progress.

Action planning will be tailored by the bilingual ONN through linguistic (i.e., action plan worksheet translation and delivery in English or Spanish), evidential (presenting evidence on the importance of comorbidity management during cancer treatment), and sociocultural strategies (i.e., integrating cultural values and religious beliefs when addressing barriers and facilitators to behavior change), as appropriate. Afterwards, the ONN will check in with the patient at his or her routine 2 and 4 month clinic visits to follow up on action plan progress, address concerns, and confirm survey completion.

Tailored survivorship action planning. After cancer treatment completion, as per UMC, the Survivorship NP will schedule a transition review appointment where he or she will review the SCP and educate patients about prevention and surveillance guidelines, long term and late effects, and recommended lifestyle modifications. After this, the ONN will meet with the patient to reinforce the SCP, and provide him or her with a referral to the PCP (to conduct a physical exam, discuss any adjustments to the comorbidity management plan that may be needed in light of cancer treatment completion, and coordinate specialty care referrals), discuss different roles and responsibilities of the oncologist and PCP post treatment, and provide the patient with hospital and community resources for cancer survivors. The ONN and patient will collaborate to develop a culturally tailored survivorship self management action plan. Afterwards, patients will complete the next scheduled assessment survey and the RA will gauge patient interest in participating in an additional optional interview within 1 month of SCP delivery. The purpose is to obtain a more in depth perspective regarding patient knowledge and understanding of the SCP, unmet needs, and experiences with comorbidity management during cancer treatment. Recruitment for the qualitative interviews will continue until we have reached 30 patients (N=15 for each study arm) or saturation has been achieved. Interviews will be conducted by phone, last 60 minutes, and be digitally recorded and transcribed. Surveillance reminders and follow up. Patients will receive reminders of upcoming surveillance visits via phone or text message to encourage adherence. The ONN will meet with patients after their oncology surveillance visits to 1) ensure ongoing care management with the PCP, 2) follow up on action plan progress, 3) answer questions, and 4) confirm survey completion. After surveillance visits with the PCP, the ONN will review progress reports and relevant test results, report them to the oncologist, and follow up by sending a memo via EPIC to request clarifications if needed. Provider Decision Support. Treatment plan and concerns. When the initial PCP referral is made, the ONN will send the PCP treatment plan summary (based on the ASCO treatment plan template) and standardized fact sheets on treatment toxicities that we will develop.

Bi directional and structured communication between oncologist and PCP. Throughout cancer treatment, the ONN will be available to answer questions from PCP staff and facilitate prompt communication between the oncologist and PCP as questions arise. Surveillance guidelines and summary of late effects. The SCP will be sent to the PCP via the EHR, along with a memo detailing surveillance guidelines, oncologist concerns related to the management of treatment toxicities and late effects, and recommendations for specialty care referrals (e.g., cardiology, nutrition, physical therapy). Clinical Information Systems. EHR enhancements. We will work with the Harris Health EPIC Information Technology (IT) group to create and streamline templates for treatment summaries and to generate standardized toxicity and concern lists to facilitate coordination of care between oncologists and PCPs. EHR generated SCP. After treatment completion, the oncologist will classify the patient as low , moderate or high risk for recurrence based on the treatment received, presence and degree of persistent therapy toxicity, presence and degree of organ dysfunction, and risk of developing serious late effects. This will be entered in the EHR and used to populate surveillance visit recommendations in the SCP.

Delivery System Redesign. OPTIMISE will adopt a risk stratified shared care model of post treatment survivorship care. As patients typically see their oncologist for surveillance 3-4 times in the first year post treatment, OPTIMISE participants will undergo a risk stratified shared care model in which a certain number of oncologist surveillance visits are replaced by PCP visits. For low risk patients, one oncologist visit will be replaced by a PCP visit. Moderate and high risk patients will receive all surveillance visits from the oncologist (none replaced). All patients will complete follow up surveys at 3, 6, and 12 months post SCP delivery in the clinic or by mail.

Linkages to Community Resources. Patients will receive resource lists linking them to healthcare and community resources at diagnosis, during treatment, and at SCP delivery. Provider interviews will elucidate opportunities for increased community linkages that will inform future scale out efforts. Healthcare Organization Support. To inform strategies to support future scale up, we will conduct interviews with providers to identify factors affecting care coordination, SCP delivery, and care transitions.

ELIGIBILITY:
Inclusion Criteria:

* For patients: 1) new diagnosis or within three months of treatment initiation for early-stage breast (I-IIIB), GI (Stage I-III), or hematologic (Stage I-III) cancer 2) treatment with standard, definitive therapies (may include one or more modalities) 3) presence of one or more chronic comorbidities (e.g., diabetes, hypertension) and/or unhealthy lifestyle behaviors (e.g., overweight/obesity, current smoker, alcohol use) that require ongoing management during cancer treatment 4) age >18 years 5) fluency in English or Spanish 6) ability to provide informed consent 7) assignment to a Harris Health oncologist and PCP who are willing to participate and will provide informed consent.

For healthcare providers: 1) Person is an oncologist or PCP who treats patients with breast, GI, or hematologic malignancies at Harris Health BT/Smith Clinic

Exclusion Criteria:

* For Patients: Significant cognitive impairment or Lack of capacity to consent For Providers: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM) | 4 month follow-up
  self-management attitudes
Instrument to measure Self-Management (IMSM) | 4 month follow-up
  self-management behaviors

SECONDARY OUTCOMES:
Function Assessment of Cancer Therapy (FACT-G) | 4 month follow-up
  Quality of life
Supportive Care Needs Survey (SCNS) | 4 month follow-up
  patient unmet needs

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Badr, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No